CLINICAL TRIAL: NCT05338229
Title: The Engineer-built System, Video-game Based Kinect Sensor in Upper Extremities Problems in Cerebral Palsy Children: Phase 2.1
Brief Title: Kinect Sensor in Cerebral Palsy Children: Phase 2.1
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocal changing due to time limitation
Sponsor: Mahidol University (Other)
Collaborators: Warakorn Charoensuk (Unknown); Apiphan Iamchaimongkol (Unknown); Tulyapruek Tawonsawatruk (Unknown)
Responsible Party: Principal Investigator, Sivaporn Vongpipatana, Assistant Professor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MURA2021/768-2.1
Record Dates: First submitted 2022-03-25; First posted 2022-04-21 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Cerebral Palsy Children; Upper Extremity Problem
Keywords: video-game; Kinect sensor; upper extremities problems; cerebral palsy; children
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- video game in CP children (pilot study) (Experimental): The cerebral palsy children will play the engineer-built system, video-game based Kinect sensor 3 times/week for 5 weeks. Each session will last for 40 minutes. The video-game Kinect sensor was developed by the researcher team.
  Interventions: Device: the engineer-built system, video-game based Kinect sensor

INTERVENTIONS:
Device: the engineer-built system, video-game based Kinect sensor — The engineer-built system, video-game based Kinect sensor was developed by the researcher team.

SUMMARY:
There are 3 phases of the study. This registration is phase 2.1.This registration will conduct a pilot study in the cerebral palsy children.

ELIGIBILITY:
Inclusion Criteria:

* Spastic cerebral palsy aged 10-15 years
* Sufficient cognitive/attention capacity to understand basic instructions
* Can cooperate with the therapist for short period of time during training
* Manual Ability Classification System (MACS) 2-3
* Zancolli classification of the affected upper extremity was grade I-II.
* Give the informed consent

Exclusion Criteria:

* Inability to understand the instruction and follow the task
* Severe comorbidities, visual or auditory impairment
* Had history of Botulinum toxin injection on the affected upper extremity for last 6 months or receive the injection during the study time
* Other treatment options planned on the affected upper extremity during the study time
* Wear daytime orthosis on the affected limb
* Zancolli classification of the affected hand was grade III.
* Got an epilepsy or convulsive condition
* Denied to give the informed consent or continue the study

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Range of Motion | before starting the intervention and after finishing the intervention within 1 week
  The range or motion of shoulder, elbow and wrist will be assessed by goniometer. The assessment will be done before starting the intervention as the baseline and then after finishing the intervention to detect change of range of motion from the the baseline. The range of motion will be reported in degrees.

SECONDARY OUTCOMES:
Box and block test | before starting the intervention and after finishing the intervention within 1 week
  The name 'box and block test' is an unabbreviated scale title. The minimum score is zero and the maximum score is infinity.
ABILHANDS-Kids | before starting the intervention and after finishing the intervention within 1 week
  The ABILHANDS-kids is the name of the test. It is not an unabbreviated name. The children will be asked the difficulty of doing their activities of daily living by using 21 questionnaires. The rating of difficulties were impossible, difficult and easy. Then the rating would be score as impossible=0, difficult=1 and easy = 2. The analysis of the score of there items will use the Rasch analysis which it is available online on http://rssandbox.iescagilly.be/~abilhand-kids-cerebral-palsy-en.html. The minimum score means a worse outcome and the maximum score means the better outcome.
EQ-5D-Y | before starting the intervention and after finishing the intervention within 1 week
  The EQ-5D-Y is a questionnaire which has 2 parts for a participant to complete. There are 5 questions asking in first part: mobility, looking after myself, doing usual activities, having pain or discomfort and feelin worried, sad or unhappy. The participant needs to rate these questions in 3 rating score: no problem, with some problem or with a lot of problem. The rating score will be coded as no problem=1, with some problem = 1 and with a lot of problem = 2. The code 11111 is the best condition and the code 33333 is the worst condition. The second part of the questionnaire is the EQ-VAS which the participants need to rate their condition on the linear scale from 0-100. The worst condition is score 0 and the best condition is score 100.Then the coding from the first part will be converted as an index value.

OTHER OUTCOMES:
patient satisfaction form | immediately after finishing the intervention
  The patient satisfaction form is about the questionnaire asking about the satisfaction of playing game in these areas: the presentation of games: the contents of game, the convenience and the outcome after playing game. The participants will rate each question in 5-likert scale: totally disagree, disagree, neutral, agree and totally agree.

CONTACTS AND LOCATIONS:
Overall Officials: Sivaporn Vongpipatana, Principal Investigator — Department of Rehabilitation Medicine, Faculty of Medicine Ramathibodi Hospital Mahidol University

IPD SHARING:
Plan to Share IPD: Yes
I plan to share the information about the result of the study with the statistician and some team members for the analysis. The sharing will not be linked to the patient identification.
Supporting Information: SAP, Analytic Code
Time Frame: within 3 months after harvesting the data

REFERENCES:
- [Background] Arneson CL, Durkin MS, Benedict RE, Kirby RS, Yeargin-Allsopp M, Van Naarden Braun K, Doernberg NS. Prevalence of cerebral palsy: Autism and Developmental Disabilities Monitoring Network, three sites, United States, 2004. Disabil Health J. 2009 Jan;2(1):45-8. doi: 10.1016/j.dhjo.2008.08.001. PMID 21122742
- [Background] Bhasin TK, Brocksen S, Avchen RN, Van Naarden Braun K. Prevalence of four developmental disabilities among children aged 8 years--Metropolitan Atlanta Developmental Disabilities Surveillance Program, 1996 and 2000. MMWR Surveill Summ. 2006 Jan 27;55(1):1-9. PMID 16437058
- [Background] Paneth N, Hong T, Korzeniewski S. The descriptive epidemiology of cerebral palsy. Clin Perinatol. 2006 Jun;33(2):251-67. doi: 10.1016/j.clp.2006.03.011. PMID 16765723
- [Background] Prevalence and characteristics of children with cerebral palsy in Europe. Dev Med Child Neurol. 2002 Sep;44(9):633-40. PMID 12227618
- [Background] Chen YP, Lee SY, Howard AM. Effect of virtual reality on upper extremity function in children with cerebral palsy: a meta-analysis. Pediatr Phys Ther. 2014 Fall;26(3):289-300. doi: 10.1097/PEP.0000000000000046. PMID 24819682
- [Background] Samia Abdel Rahman, Abdel Rahman, Afaf A. Shaheen. Virtual Reality Use in Motor Rehabilitation of Neurological Disorders: A Systematic Review. Middle-East Journal of Scientific Research; 7 (1): 63-70.
- [Background] Chen YP, Kang LJ, Chuang TY, Doong JL, Lee SJ, Tsai MW, Jeng SF, Sung WH. Use of virtual reality to improve upper-extremity control in children with cerebral palsy: a single-subject design. Phys Ther. 2007 Nov;87(11):1441-57. doi: 10.2522/ptj.20060062. Epub 2007 Sep 25. PMID 17895352
- [Background] Green D, Wilson PH. Use of virtual reality in rehabilitation of movement in children with hemiplegia--a multiple case study evaluation. Disabil Rehabil. 2012;34(7):593-604. doi: 10.3109/09638288.2011.613520. Epub 2011 Oct 6. PMID 21978233
- [Background] Pruksananonda C. Cerebral Palsy. In: Prasongjean P, editor. Cerebral Palsy Disease. Bangkok: Chulalongkorn University Printing House; 2010. p. 1-3.